CLINICAL TRIAL: NCT03943888
Title: Pharmacokinetic-pharmacodynamic Analysis of Reversal of Rocuronium-induced Neuromuscular Blockade by Sugammadex in Children
Brief Title: Pharmacokinetic-pharmacodynamic Analysis of Sugammadex in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Hee-Soo Kim, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1904-149-1029
Record Dates: First submitted 2019-05-06; First posted 2019-05-09 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Anesthesia, General; Neuromuscular Blockade
Keywords: sugammadex; pharmacokinetics; pharmacodynamics; pediatric anesthesia
MeSH Terms: interventions — Sugammadex; Atropine; Neostigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Sugammadex 2mg (Experimental): Administer 2mg/kg of sugammadex 15 minutes after rocuronium administration
  Interventions: Drug: Sugammadex Injection 2mg/kg
- Sugammadex 4mg (Experimental): Administer 4mg/kg of sugammadex 15 minutes after rocuronium administration
  Interventions: Drug: Sugammadex Injection 4mg/kg
- Sugammadex 8mg (Experimental): Administer 8mg/kg of sugammadex 15 minutes after rocuronium administration
  Interventions: Drug: Sugammadex Injection 8mg/kg
- Conventional reversal (Active Comparator): Administer conventional neuromuscular reversal agent (0.02mg/kg of atropine and 0.03mg/kg of neostigmine) 15 minutes after rocuronium administration
  Interventions: Drug: Neuromuscular reversal agent injection

INTERVENTIONS:
Drug: Sugammadex Injection 2mg/kg — Intravenous injection of 2mg/kg of sugammadex sodium 15 minutes after rocuronium administration
  Other Names: Bridion 2mg/kg
  Arms: Sugammadex 2mg
Drug: Sugammadex Injection 4mg/kg — Intravenous injection of 4mg/kg of sugammadex sodium 15 minutes after rocuronium administration
  Other Names: Bridion 4mg/kg
  Arms: Sugammadex 4mg
Drug: Sugammadex Injection 8mg/kg — Intravenous injection of 8mg/kg of sugammadex sodium 15 minutes after rocuronium administration
  Other Names: Bridion 8mg/kg
  Arms: Sugammadex 8mg
Drug: Neuromuscular reversal agent injection — Intravenous injection of 0.02mg/kg of atropine and 0.03mg/kg of neostigmine
  Other Names: Atropine and neostigmine
  Arms: Conventional reversal

SUMMARY:
This study administers sugammadex sodium to pediatric patients under general anesthesia with rocuronium. Pharmacokinetic and pharmacodynamic analysis are performed based on plasma concentration of sugammadex sodium and monitoring of neuromuscular blockade.

DETAILED DESCRIPTION:
This study enrolls pediatric patients undergoing surgery under general anesthesia with need for early reversal of neuromuscular blockade, aged between 2 and 18 years old.

After routine anesthetic induction with 1% propofol and 0.6mg/kg of rocuronium, maintenance of anesthesia with total intravenous anesthesia is commenced. 15 minutes after rocuronium administration, 2 or 4 or 8mg/kg of sugammadex sodium or conventional neuromuscular reversal agent is administered according to randomization table.

For neuromuscular monitoring, train-of-four (TOF) count and T4/T1 ratio are monitored, with recording of the time to recovery of the T4/T1 ratio to 0.7, 0.8 and 0.9.

For pharmacokinetic analysis, patient blood sample is obtained before / 2 min after rocuronium administration, before / 2min / 5min / 15min / 60min / 120min / 240min / 480min after sugammadex administration. Plasma concentration of rocuronium and sugammadex sodium are analyzed via high-performance liquid chromatography with mass spectrometric detection.

ELIGIBILITY:
Inclusion Criteria: All of below

* Pediatric patients undergoing surgery under general anesthesia with requirement of early reversal of neuromuscular blockade
* Aged between 2 and 17
* American Society of Anesthesiologists Physical Status Classification 1 and 2

Exclusion Criteria: Any of below

* One or more legal guardian declines to enroll in the study
* History of hypersensitivity to any anesthetic agents including rocuronium
* Presence of underlying cardiovascular or genitourinary disease
* Under usage of neuromuscular blocking agents before surgery
* Under usage of drugs influencing the effect of neuromuscular blocking agents
* History of malignant hyperthermia
* Anticipation of massive hemorrhage during surgery

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, M.D, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gijsenbergh F, Ramael S, Houwing N, van Iersel T. First human exposure of Org 25969, a novel agent to reverse the action of rocuronium bromide. Anesthesiology. 2005 Oct;103(4):695-703. doi: 10.1097/00000542-200510000-00007. PMID 16192761
- [Background] Sorgenfrei IF, Norrild K, Larsen PB, Stensballe J, Ostergaard D, Prins ME, Viby-Mogensen J. Reversal of rocuronium-induced neuromuscular block by the selective relaxant binding agent sugammadex: a dose-finding and safety study. Anesthesiology. 2006 Apr;104(4):667-74. doi: 10.1097/00000542-200604000-00009. PMID 16571960
- [Background] Sparr HJ, Vermeyen KM, Beaufort AM, Rietbergen H, Proost JH, Saldien V, Velik-Salchner C, Wierda JM. Early reversal of profound rocuronium-induced neuromuscular blockade by sugammadex in a randomized multicenter study: efficacy, safety, and pharmacokinetics. Anesthesiology. 2007 May;106(5):935-43. doi: 10.1097/01.anes.0000265152.78943.74. PMID 17457124
- [Background] Ploeger BA, Smeets J, Strougo A, Drenth HJ, Ruigt G, Houwing N, Danhof M. Pharmacokinetic-pharmacodynamic model for the reversal of neuromuscular blockade by sugammadex. Anesthesiology. 2009 Jan;110(1):95-105. doi: 10.1097/ALN.0b013e318190bc32. PMID 19104176
- [Background] Won YJ, Lim BG, Lee DK, Kim H, Kong MH, Lee IO. Sugammadex for reversal of rocuronium-induced neuromuscular blockade in pediatric patients: A systematic review and meta-analysis. Medicine (Baltimore). 2016 Aug;95(34):e4678. doi: 10.1097/MD.0000000000004678. PMID 27559972

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugammadex 2mg | Sugammadex 4mg | Sugammadex 8mg | Conventional Reversal
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex 2mg | Sugammadex 4mg | Sugammadex 8mg | Conventional Reversal | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 10 | 10 | 40
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 6.5 [3.5 to 15] | 10 [3.7 to 16] | 6 [3.5 to 15] | 8.5 [4 to 13] | 7 [3.5 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 4 | 5 | 19
  Male | 6 | 4 | 6 | 5 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 10 | 10 | 10 | 10 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 10 | 10 | 10 | 10 | 40
Type of surgery [Count of Participants; unit: Participants]
  Brain | 6 | 4 | 7 | 10 | 27
  Spine | 4 | 6 | 3 | 0 | 13

OUTCOME MEASURES:

1. Primary Outcome: Neuromuscular Recovery
Description: Time to recovery of train-of-four T4/T1 ratio to 90% after sugammadex sodium or neuromuscular reversal agent administration up to 30 minutes to 1 hour.
Time Frame: up to 30 minutes to 1 hour
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex 2mg | Sugammadex 4mg | Sugammadex 8mg | Conventional Reversal
Number analyzed (Participants) | 10 | 10 | 10 | 10
Minutes | 5.7 (4.7) | 3.1 (1.0) | 1.1 (1.0) | 43.7 (28.2)

2. Secondary Outcome: Plasma Concentrations
Description: Plasma concentrations of rocuronium and sugammadex sodium
Time Frame: From anesthetic induction to 480 minutes after sugammadex administration
Population: Cmax of sugammadex and rocuronium
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Sugammadex 2mg | Sugammadex 4mg | Sugammadex 8mg | Conventional Reversal
Number analyzed (Participants) | 10 | 10 | 10 | 10
mcg/mL
  Sugammadex: number analyzed (Participants) | 10 | 10 | 10 | 0
  Sugammadex | 28.5 (9.6) | 58.2 (12.5) | 118.9 (13) |
  Rocuronium: number analyzed (Participants) | 9 | 9 | 9 | 10
  Rocuronium | 5.3 (1.9) | 8.0 (2.1) | 5.4 (3) | 6.8 (3.1)

ADVERSE EVENTS:
Time Frame: From the start of anesthesia to 24 hours after the end of surgery.
Description: No mortality, serious adverse event, adverse event related to study drug were observed during the study.
Arm/Group | Sugammadex 2mg | Sugammadex 4mg | Sugammadex 8mg | Conventional Reversal
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03943888/Prot_SAP_000.pdf